CLINICAL TRIAL: NCT01835353
Title: High (100mg) Versus Standard (60mg) Loading Dose of Prasugrel in Patients With ST-elevation Myocardial Infarction (STEMI), Undergoing Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-13
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Platelet Reactivity
Keywords: prasugrel; ST elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel 100mg loading dose (Experimental): Prasugrel 100mg loading dose
  Interventions: Drug: Prasugrel 100mg loading dose
- Prasugrel 60mg loading dose (Active Comparator)
  Interventions: Drug: Prasugrel 60mg loading dose

INTERVENTIONS:
Drug: Prasugrel 100mg loading dose
  Arms: Prasugrel 100mg loading dose
Drug: Prasugrel 60mg loading dose — Prasugrel 60mg loading dose
  Arms: Prasugrel 60mg loading dose

SUMMARY:
This is a prospective, multi-center, non-randomized, controlled study in 2 sequential groups of P2Y12 inhibitor-naive consecutive STEMI patients undergoing primary PCI. Following aspirin 325 mg LD, patients will receive 60 mg or 100 mg of prasugrel, respectively. Platelet reactivity (PR)will be assessed at Hour 0 (before prasugrel's administration immediately prior to PCI) and at Hours 0.5, 1, 2, 4 thereafter. Platelet function testing (in PRU) will be performed with the VerifyNow (Accumetrics Inc., San Diego, CA, USA) P2Y12 function assay.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction
* Pain onset <12 hours
* Age >18 and <75 years
* Written informed consent

Exclusion Criteria:

* history of stroke/transient ischemic attack
* oral anticoagulation
* hemodynamic instability
* platelet count <100000/μL
* hematocrit <30%
* creatinine clearance <30 ml/min
* severe hepatic dysfunction
* active bleeding
* weight <60 Kg
* periprocedural IIb/IIIa inhibitor administration

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity in Platelet reactivity units (PRU) at Hour 2 | 2 hours
  Platelet reactivity in Platelet reactivity units (PRU) 2 hours post randomization

SECONDARY OUTCOMES:
Platelet reactivity in platelet reactivity units (PRU)at hour 1 | 1 hour
  Platelet reactivity in platelet reactivity units (PRU)1 hour post randomization
Platelet reactivity in platelet reactivity units (PRU)at hour 0.5 | 0.5 hours
  Platelet reactivity in platelet reactivity units (PRU)0.5 hour post randomization
Platelet reactivity in platelet reactivity units (PRU)at hour 4 | 4 hours
  Platelet reactivity in platelet reactivity units (PRU)4 hours post randomization
High platelet reactivity rate (208 PRU threshold) at 0.5 hour | 0.5 hour
  High platelet reactivity rate (208 PRU threshold) 0.5 hour post randomization
High platelet reactivity rate (208 PRU threshold) at 1 hour | 1 hour
  High platelet reactivity rate (208 PRU threshold) 1 hour post randomization
High platelet reactivity rate (208 PRU threshold) at 2 hour | 2 hours
  High platelet reactivity rate (208 PRU threshold) 2 hours post randomization
High platelet reactivity rate (208 PRU threshold) at 4 hour | 4 hours
  High platelet reactivity rate (208 PRU threshold) 4 hours post randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Dimitrios Alexopoulos, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Makris G, Xanthopoulou I, Patsilinakos S, Deftereos S, Gkizas V, Perperis A, Karanikas S, Angelidis C, Tsigkas G, Koutsogiannis N, Hahalis G, Davlouros P. Onset of antiplatelet action with high (100 mg) versus standard (60 mg) loading dose of prasugrel in patients with ST-segment-elevation myocardial infarction undergoing primary percutaneous coronary intervention: pharmacodynamic study. Circ Cardiovasc Interv. 2014 Apr;7(2):233-9. doi: 10.1161/CIRCINTERVENTIONS.113.001118. Epub 2014 Mar 25. PMID 24668226